CLINICAL TRIAL: NCT04671186
Title: Role of Probiotics in Treatment of Pediatric Nonalcoholic Fatty Liver Disease (NAFLD) Patients by Assessing With Fibroscan
Brief Title: Role of Probiotics in Treatment of Pediatric NAFLD Patients by Assessing With Fibroscan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-0198
Record Dates: First submitted 2020-09-01; First posted 2020-12-17 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Non-Alcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Intervention Model Description: Participants will be blindly randomized at Visit 1 into one of two groups (probiotic or placebo). Probiotic group will receive Lactobacillus rhamnosus strain GG one capsule oral daily (10 billion CFU/day) and the other group receive placebo oral capsule daily throughout the study. All participants in either group will undergo: Life style modification as per NASPGHAN NAFLD guidelines. Fibroscan assessing CAP and TE score once every 3 month until the end of study. Monitoring ALT every 3 months until end of study as per standard of care guidelines.Collection of stool sample to be sent for microbiome analysis at the time of diagnosis, 3 months and 6 months (end of the study). Secondary variables collected, Age, Gender, Race, BMI, Fibroscan probe.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants will be blindly randomized at baseline (Visit 1) into one of two groups: probiotic or placebo. Investigators are to be blinded as well
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic group (Experimental): Probiotic group will receive Lactobacillus rhamnosus strain GG one capsule oral daily (10 billion CFU/day) throughout the study
  Interventions: Dietary Supplement: Culturelle (Lactobacillus rhamnosus strain GG)
- Placebo Group (Placebo Comparator): Placebo group is to receive placebo oral capsule daily throughout the study.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Culturelle (Lactobacillus rhamnosus strain GG) — Culturelle probiotics are typically sold over the counter as dietary supplements Probiotics group will take 1 capsule of probiotics orally once daily
  Arms: Probiotic group
Other: Placebo — Placebo group will take 1 capsule of placebo orally once daily
  Arms: Placebo Group

SUMMARY:
The goal of this study is to evaluate the role of probiotics in the treatment of pediatric NAFLD by evaluating for steatosis and fibrosis with a Fibroscan machine. This will be done by performing a fibroscan during each visit and comparing patients' ALT at various intervals. This is an important study as current pediatric guidelines only recommend lifestyle modifications for the treatment of NAFLD and the use of ALT and sonogram to assess improvement as standard of care. Investigators hypothesized that treatment with a probiotic will demonstrate an improvement in NAFLD as assessed by a fibroscan of liver which is good for the monitoring of steatosis and fibrosis. Additionally, analysis of fecal microbiome results may offer insight into targeted therapy in the future.

DETAILED DESCRIPTION:
The goal/objective of this study is to evaluate the role of probiotics in the treatment of NAFLD by assessing with fibroscan in both newly diagnosed and known pediatric patients with NAFLD. This will be done by performing a fibroscan during each visit and comparing patient ALT and fecal microbiome at various intervals.

The primary endpoint is to assess the effect of probiotic treatment in liver steatosis and fibrosis by assessing with fibroscan using CAP score and TE staging. The higher the CAP score (S1, S2, S3) so worse the steatosis. TE staging (F0-F4), higher the staging indicates worsening of fibrosis.

Secondary endpoints include:

* The rate of decline of ALT over 3 month time interval and through whole study starting at initial diagnosis.
* The rate of decrease in hepatic steatosis and BMI

This study will target pediatric patients with NAFLD. Participants will be new and previously diagnosed NAFLD patients between the ages of 5 years and 18 years.

This is single center study. Investigators will enroll patients from The Division of Pediatric Gastroenterology, Liver Disease and Nutrition.

Participants will be blindly randomized into one of two groups: probiotic or placebo.

Investigators expect the study to run for 1 year from 09/15/2020 to 09/14/2021. Investigators will enroll patients over a 6 month period. After randomization into two separate groups (probiotic vs placebo), Investigators plan to collect data for the subsequent 6 months following enrollment.

ELIGIBILITY:
Inclusion Criteria:

* This study will target pediatric patients with NAFLD. Participants will be new and previously diagnosed NAFLD patients between the ages of 5 years and 18 years. Diagnosis must be made by elevated serum ALT (two times above the sex specific upper limit of normal) and a sonogram consistent with steatosis

Exclusion Criteria:

* Exclusion criteria for both groups

  * Concomitant underlying liver disease such as but not limited to autoimmune hepatitis
  * Concomitant infectious hepatitis
  * Medication use of steroids, methotrexate, metformin, and therapeutic dose of Vit. E
  * Recent antibiotic use in last 4 weeks
  * Clinically significant weight loss (at least 5% reduction in weight from baseline level [18]) on follow up NAFLD patients who were on life style modification intervention
  * Cirrhosis (Fibroscan score ≥14.0)>

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 47 (Actual)
Dates: Start 2020-09-07 (Actual); Primary Completion 2021-09-06 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
The role of probiotics in the treatment of pediatric NAFLD by evaluating for steatosis with a Fibroscan machine. | One year
  The primary endpoint/outcome assesses the effect of probiotic treatment in liver steatosis by assessing with fibroscan using CAP score.
The role of probiotics in the treatment of pediatric NAFLD by evaluating for fibrosis with a Fibroscan machine. | One year
  The primary endpoint/outcome assesses the effect of probiotic treatment in liver fibrosis by assessing with fibroscan using TE staging.

SECONDARY OUTCOMES:
Rate of decline in ALT. | One year
  The rate of decline of ALT over 3 month time interval and through whole study starting at initial diagnosis.
Change in fecal microbiome | One year
  Compare changes in stool microbiome
Decrease in BMI | One year
  The rate of change in hepatic steatosis with change in BMI

CONTACTS AND LOCATIONS:
Overall Officials: Shari Sheflin-Findling, Principal Investigator — Cohen Children's Medical Center
Locations (1):
- Cohen Children's Medical Center, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wong RJ, Aguilar M, Cheung R, Perumpail RB, Harrison SA, Younossi ZM, Ahmed A. Nonalcoholic steatohepatitis is the second leading etiology of liver disease among adults awaiting liver transplantation in the United States. Gastroenterology. 2015 Mar;148(3):547-55. doi: 10.1053/j.gastro.2014.11.039. Epub 2014 Nov 25. PMID 25461851
- [Background] Alisi A, Manco M, Vania A, Nobili V. Pediatric nonalcoholic fatty liver disease in 2009. J Pediatr. 2009 Oct;155(4):469-74. doi: 10.1016/j.jpeds.2009.06.014. No abstract available. PMID 19772998
- [Background] Paolella G, Mandato C, Pierri L, Poeta M, Di Stasi M, Vajro P. Gut-liver axis and probiotics: their role in non-alcoholic fatty liver disease. World J Gastroenterol. 2014 Nov 14;20(42):15518-31. doi: 10.3748/wjg.v20.i42.15518. PMID 25400436
- [Background] Vos MB, Abrams SH, Barlow SE, Caprio S, Daniels SR, Kohli R, Mouzaki M, Sathya P, Schwimmer JB, Sundaram SS, Xanthakos SA. NASPGHAN Clinical Practice Guideline for the Diagnosis and Treatment of Nonalcoholic Fatty Liver Disease in Children: Recommendations from the Expert Committee on NAFLD (ECON) and the North American Society of Pediatric Gastroenterology, Hepatology and Nutrition (NASPGHAN). J Pediatr Gastroenterol Nutr. 2017 Feb;64(2):319-334. doi: 10.1097/MPG.0000000000001482. PMID 28107283
- [Background] Comparison of Controlled Attenuation Parameter and Liver Biopsy to Assess Hepatic Steatosis in Pediatric PatientsAuthor links open overlay panel NiravK.DesaiMD1,SarahHarneyBA1,RoshanRazaMD1,AlyaaAlIbraheemiMD2, NickShillingfordMD2, Paul D.MitchellMS3, Maureen M.JonasMD1
- [Background] Schwimmer JB, Newton KP, Awai HI, Choi LJ, Garcia MA, Ellis LL, Vanderwall K, Fontanesi J. Paediatric gastroenterology evaluation of overweight and obese children referred from primary care for suspected non-alcoholic fatty liver disease. Aliment Pharmacol Ther. 2013 Nov;38(10):1267-77. doi: 10.1111/apt.12518. Epub 2013 Oct 1. PMID 24117728
- [Background] Draijer L, Benninga M, Koot B. Pediatric NAFLD: an overview and recent developments in diagnostics and treatment. Expert Rev Gastroenterol Hepatol. 2019 May;13(5):447-461. doi: 10.1080/17474124.2019.1595589. Epub 2019 Apr 4. PMID 30875479
- [Background] Leung C, Rivera L, Furness JB, Angus PW. The role of the gut microbiota in NAFLD. Nat Rev Gastroenterol Hepatol. 2016 Jul;13(7):412-25. doi: 10.1038/nrgastro.2016.85. Epub 2016 Jun 8. PMID 27273168
- [Background] Lau E, Carvalho D, Freitas P. Gut Microbiota: Association with NAFLD and Metabolic Disturbances. Biomed Res Int. 2015;2015:979515. doi: 10.1155/2015/979515. Epub 2015 May 19. PMID 26090468
- [Background] Ley RE, Backhed F, Turnbaugh P, Lozupone CA, Knight RD, Gordon JI. Obesity alters gut microbial ecology. Proc Natl Acad Sci U S A. 2005 Aug 2;102(31):11070-5. doi: 10.1073/pnas.0504978102. Epub 2005 Jul 20. PMID 16033867
- [Background] Ley RE, Peterson DA, Gordon JI. Ecological and evolutionary forces shaping microbial diversity in the human intestine. Cell. 2006 Feb 24;124(4):837-48. doi: 10.1016/j.cell.2006.02.017. PMID 16497592
- [Background] Henao-Mejia J, Elinav E, Jin C, Hao L, Mehal WZ, Strowig T, Thaiss CA, Kau AL, Eisenbarth SC, Jurczak MJ, Camporez JP, Shulman GI, Gordon JI, Hoffman HM, Flavell RA. Inflammasome-mediated dysbiosis regulates progression of NAFLD and obesity. Nature. 2012 Feb 1;482(7384):179-85. doi: 10.1038/nature10809. PMID 22297845
- [Background] Mouzaki M, Comelli EM, Arendt BM, Bonengel J, Fung SK, Fischer SE, McGilvray ID, Allard JP. Intestinal microbiota in patients with nonalcoholic fatty liver disease. Hepatology. 2013 Jul;58(1):120-7. doi: 10.1002/hep.26319. Epub 2013 May 14. PMID 23401313
- [Background] Le Roy T, Llopis M, Lepage P, Bruneau A, Rabot S, Bevilacqua C, Martin P, Philippe C, Walker F, Bado A, Perlemuter G, Cassard-Doulcier AM, Gerard P. Intestinal microbiota determines development of non-alcoholic fatty liver disease in mice. Gut. 2013 Dec;62(12):1787-94. doi: 10.1136/gutjnl-2012-303816. Epub 2012 Nov 29. PMID 23197411
- [Background] Alisi A, Bedogni G, Baviera G, Giorgio V, Porro E, Paris C, Giammaria P, Reali L, Anania F, Nobili V. Randomised clinical trial: The beneficial effects of VSL#3 in obese children with non-alcoholic steatohepatitis. Aliment Pharmacol Ther. 2014 Jun;39(11):1276-85. doi: 10.1111/apt.12758. Epub 2014 Apr 16. PMID 24738701
- [Background] Vajro P, Mandato C, Licenziati MR, Franzese A, Vitale DF, Lenta S, Caropreso M, Vallone G, Meli R. Effects of Lactobacillus rhamnosus strain GG in pediatric obesity-related liver disease. J Pediatr Gastroenterol Nutr. 2011 Jun;52(6):740-3. doi: 10.1097/MPG.0b013e31821f9b85. PMID 21505361
- [Background] Ferolla SM, Armiliato GN, Couto CA, Ferrari TC. Probiotics as a complementary therapeutic approach in nonalcoholic fatty liver disease. World J Hepatol. 2015 Mar 27;7(3):559-65. doi: 10.4254/wjh.v7.i3.559. PMID 25848479
- [Background] Swift DL, Johannsen NM, Lavie CJ, Earnest CP, Blair SN, Church TS. Effects of clinically significant weight loss with exercise training on insulin resistance and cardiometabolic adaptations. Obesity (Silver Spring). 2016 Apr;24(4):812-9. doi: 10.1002/oby.21404. Epub 2016 Mar 3. PMID 26935138
- [Background] Patton HM, Yates K, Unalp-Arida A, Behling CA, Huang TT, Rosenthal P, Sanyal AJ, Schwimmer JB, Lavine JE. Association between metabolic syndrome and liver histology among children with nonalcoholic Fatty liver disease. Am J Gastroenterol. 2010 Sep;105(9):2093-102. doi: 10.1038/ajg.2010.152. Epub 2010 Apr 6. PMID 20372110
- [Background] Fusillo S, Rudolph B. Nonalcoholic fatty liver disease. Pediatr Rev. 2015 May;36(5):198-205; quiz 206. doi: 10.1542/pir.36-5-198. PMID 25934909
- [Background] Awai HI, Newton KP, Sirlin CB, Behling C, Schwimmer JB. Evidence and recommendations for imaging liver fat in children, based on systematic review. Clin Gastroenterol Hepatol. 2014 May;12(5):765-73. doi: 10.1016/j.cgh.2013.09.050. Epub 2013 Sep 30. PMID 24090729

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04671186/Prot_SAP_000.pdf
  • Informed Consent Form (2020-04-21): https://cdn.clinicaltrials.gov/large-docs/86/NCT04671186/ICF_001.pdf